CLINICAL TRIAL: NCT03252873
Title: INVESTIGATION THE FACTORS AFFECTING THE ADHERENCE TO THE OUTPATIENT PULMONARY REHABILITATION PROGRAM IN COPD
Brief Title: THE FACTORS AFFECTING THE ADHERENCE TO THE PULMONARY REHABILITATION PROGRAM IN COPD
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof., Izmir Katip Celebi University
Other Study IDs: IzmirKCU2
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: COPD
Keywords: adherence; pulmonary rehabilitation; copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators will compare the factors affecting the adherence to the outpatient pulmonary rehabilitation program in COPD patients

DETAILED DESCRIPTION:
Patients were referred to the Pulmonary Rehabilitation Unit and were recommended to participate in the exercise program by a team of experts included in this study.

Demographic and clinical characteristics of patients were recorded before the pulmonary rehabilitation program. All cases were evaluated by pulmonary function test, arterial blood gas analysis, six minute walking test, MMRC Dyspnea Scale. Causes that prevented program adaptation of those who did not participate in the program or who left the program were questioned. Patients completing the eight-week PR program will compare with those who did not complete the program or who did not start the program at the recommended time.

ELIGIBILITY:
Inclusion Criteria: COPD Patients referred to the outpatient pulmonary rehabilitation unit -

Exclusion Criteria: To be unvolunteer

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COPD patients refered to the pulmonary rehabilitation unit.
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | 15 minutes
  FEV1 (%) FEV1 /FVC TLCO (%) FEV1 (%), FEV1 /FVC, TLCO (%)

SECONDARY OUTCOMES:
Blood Gase Analysis | 5 minutes
  PAO2, PaCO2, SaO2
Six minute walk test | 10 minutes
  walking distance
MMRC Dyspnea Scale | 5 minutes
  1-5
SGRQ Questionnaire | 20 minutes
  Symptom-Activity-Impact- Total
HAD Questionnaire | 15 minutes
  Anxiety- Depression score